CLINICAL TRIAL: NCT06422572
Title: The Role of Tissue Kallikrein - Bradykinin System Targeting the Protection of Neurovascular Units in Ischemic Areas of Stroke
Brief Title: Tissue Kallikrein Protect Against Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Qin Zhang (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Qin Zhang, PROFESSOR, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202303109
Record Dates: First submitted 2024-05-07; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2023-03

CONDITIONS: Stroke, Ischemic
Keywords: Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Part of the sample consisted of 1210 stroke controls and 905 coronary heart disease controls enrolled from December 2000 to November 2001 in the previous study. The other part comes from 6,487 cases of community population in Rizhao area from May to August 2010.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population without stroke: 1. Control population in a case-controlled study of prior stroke ;
  2. Control population in a case-controlled study of preexisting coronary heart disease;
  3. Population in previous community cross-sectional studies .
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The results of previous studies were used to assess the causal association between TK levels and stroke occurrence at 5 and 12 years of follow-up, respectively.

DETAILED DESCRIPTION:
Analyze the data of a 5-year follow-up on 2115 control individuals from the case-control study of the previous research. We completed the 5-year follow-up on this group in 2016 (whether they had a stroke, whether they are alive, and the cause of death).

Conduct a 12-year follow-up on 6487 community individuals from the previous study (whether they had a stroke within 12 years, whether they are alive, and the cause of death). We collaborated with the hospital platform's computer center to conduct follow-up through AI questionnaire surveys, followed by supplementing AI questionnaire data with telephone questionnaire surveys for those lost to follow-up.

Utilize R language R Studio 4.11 for statistical analysis and plotting. Evaluate the distribution of TK levels in the control group and its relationship with the 10-year predicted risk of stroke and the predictive role for stroke events within 5 years.

Evaluate the distribution of TK levels in the community group and its relationship with the 10-year predicted risk of stroke and the predictive role for stroke events within 12 years.

ELIGIBILITY:
Inclusion Criteria:

* 1) Control population in the previous stroke case-control study;
* 2) The CHD case-control population in the previous study;
* 3) The population in the community cross-sectional study of the previous study.

Exclusion Criteria:

* Stroke patient

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Control population in the previous stroke case-control study;
  2. The CHD case-control population in the previous study;
  3. The population in the community cross-sectional study of the previous study.
Sampling Method: Probability Sample
Enrollment: 8602 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Stroke | 5 years
  The primary outcome measure will be the occurrence of stroke during the 5-year follow-up period. Stroke events will be assessed and recorded based on predetermined diagnostic criteria, such as clinical symptoms, imaging findings, and/or medical records review. The data will be aggregated and reported as the total number of stroke cases observed in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: QIN Zhang, phd, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China